CLINICAL TRIAL: NCT05786872
Title: Efficacy and Safety of Dual-target Deep Brain Stimulation for Treatment-resistant Alcohol Use Disorder: a Multi-center, Single Arm, Prospective, Open-label, Extendable Study
Brief Title: Efficacy and Safety of Dual-target DBS for Treatment-resistant Alcohol Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Central South University (Other); Huashan Hospital (Other); Shanghai 6th People's Hospital (Other); SceneRay Corporation, Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MZhao-012
Record Dates: First submitted 2023-02-26; First posted 2023-03-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-01

CONDITIONS: Alcohol Use Disorder; Deep Brain Stimulation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dual-target deep brain stimulation (Experimental): This is a single arm, prospective, open label clinical study, participants who fit inclusion/exclusion standards, completed physical anti-addiction treatments and surgical implantation standard will start DBS system stimulation and adjust parameters after 10-14 days of implantation. Then after stimulation for 9-32 weeks, they will be evaluated for treatment efficacies. This study is extendable, with agreements from participants, long term efficacy and safety follow-up study will be performed after 32 weeks ± 7 days of following, once every 2-3 months.
  Interventions: Device: dual-target deep brain stimulation

INTERVENTIONS:
Device: dual-target deep brain stimulation — DBS electrodes will be implanted into the ALIC and the NAcc, electric stimulation of those areas are used to treat alcohol use disorder and to evaluate the efficacy and safety of DBS system.

SUMMARY:
This is a multi-center, single arm, prospective, open-label, extendable study for the efficacy and safety of dual-target deep brain stimulation for treatment-resistant alcohol use disorder.

DETAILED DESCRIPTION:
Total of 12 subjects from two centers ( Shanghai Mental Health Center and The Second Xiangya Hospital of Central South University ) who fit inclusion and exclusion criteria are recruited to undergo neurosurgical implantation of dual-target Deep Brain Stimulation (DBS) in bilateral nucleus accumbens (NAcc) and anterior limb of internal capsule (ALIC) on a certain date, the DBS system will be turned on for stimulation and parameters adjusted 10-14 days after implantation, treatment purposes are evaluated after DBS system has been turned on for 9-32 weeks. Primary efficacy is evaluated by major alcohol consumption rate, uncontrolled alcohol consumption days, maximum consecutive alcohol suspension days. Safety is evaluated by adverse events (AE) and device related AE, serious adverse events (SAE) and device related SAE, device deficiencies (DD) and device malfunction, physical examination and vital signs, laboratory examination, ECG, imageological examination, scale evaluation and early drop out ratio due to AE.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old, no limit on sex.
* Qualifies DSM-5 definition of alcohol use diagnosis, at least more than 4 terms.
* Course of alcohol use disorder ≥ 3 years.
* Tried to quit drinking (de-addiction treatment under medical conditions, quit drinking by oneself, quit drinking each time ≥ 1 week) but failed ≥ 3 times.
* Patient and relatives agree to accept systemic treatment of this study and sign Informed Consent Form after study purpose, content, expected treatment and risk etc. are fully explained and understood.

Exclusion Criteria:

* Patients who qualify DSM-5 serious mental disorder diagnosis standard (e.g. Schizophrenia spectrum, depression disorder, biphasic or related disorder, etc. )
* Patients who have other substance (tobacco excluded) abuse.
* During screening period, answered 'yes' on question 4 or 5 in suicide intention term from Columbia-Suicide Severity Rating Scale, or had significant suicide intentions in the past 3 months, or patients who are considered by researchers to have suicide or violence risks.

  4. Patients who have serious or unstable cardiovascular, respiratory, liver, kidney, hematological, endocrine, nervous system or other systemic diseases.
* Patients who have implanted cochlear, pacemaker, cardiac defibrillator, single-sided or double-sided products of the same category, or the investigator evaluates patients have done surgeries within 6 months that can affect this study.
* HIV positive patients.
* Woman at pregnant or lactation period, or childbearing age woman test positive for HCG/urine pregnancy check; or patients who can't take effective contraception measures during trial; or patients who plan to be/make pregnant 3 months after the trial starts.
* Patients who are participating other pharmaceutical or medical device clinical trials or have participated one in the past 3 months.
* Patients who are considered unsuitable by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Major alcohol use rate | 24 weeks
  Calculation formula: 'major alcohol use' times / 56 (total observation times) * 100%
Cumulated uncontrolled alcohol use days | 24 weeks
  1. Definition: more than 3 times consecutive alcohol use (random draw) ≥ 5 standard cups
  2. One time uncontrolled alcohol use days: e.g. 3 times consecutive follow-up results ≥ 5 standard cups, fourth time < 5 standard cups, then uncontrolled alcohol use days is 3 * 3 = 9 days
  3. Cumulated uncontrolled alcohol use days: Total days of all uncontrolled alcohol use days throughout 24 weeks
Maximum consecutive alcohol suspension days | 24 weeks
  a) Marked as maximum days of 'Constant alcohol suspension' b) Note: i. Major alcohol use standard: Blow test positive and reported ≥ 5 standard cups daily over the past 3 days. 1 standard cup = 10g of pure alcohol.
  ii. Minor alcohol use standard: No matter blow test is positive or not, alcohol use is reported over past 3 days but less than 5 standard cups.
  iii. Constant alcohol suspension standard: Blow test negative and no alcohol use reported over past 3 days.

SECONDARY OUTCOMES:
Alcohol use volume | 24 weeks
  9-32 weeks after stimulation, change in monthly average alcohol use volume compared to baseline. (Record in every follow-up according to participants. Record alcohol type, amount and experience when drinking throughout 9-32 weeks after stimulation. Increased value implies worse result and reduce of alcohol use volume indicates improvement.
Cumulated alcohol suspension days | 24 weeks
  total value of 'Constant alcohol suspension' days after 9-32 weeks of stimulation.
Subjective alcohol urge | At 12, 20 and 32 weeks of stimulation
  Change in alcohol urge Visual Analogue Score compared to baseline. ( 0 is no urge, 10 is extreme urge)
Alcohol abstinence | At 12, 20 and 32 weeks of stimulation
  Change in CIWA-Ar score compared to baseline.
Sleep condition | At 12, 20 and 32 weeks of stimulation
  Pittsburgh Sleep Quality Index score compared to baseline.
Emotion condition | At 12, 20 and 32 weeks of stimulation
  Hamilton Anxiety Scale-17 and Hamilton Depression Scale score compared to baseline.
Social functions | At 12, 20 and 32 weeks of stimulation
  SDSS score compared to baseline.

OTHER OUTCOMES:
Brain electrophysiology study（electroencephalogram） | Before stimulation and parameter optimization period(1-8 weeks after stimulation)
  Electroencephalographic rhythms (theta and beta) were recorded. And theta/beta ratio was compared to before stimulation
Brain electrophysiology study（Local Field Potentials） | Before stimulation and parameter optimization period(1-8 weeks after stimulation)
  Electrical signal strength was compared to before stimulation
PET-CT | Before DBS implant, after 6 months of implant.
  Before DBS implant, use Positron Emission Topography (PET) technology to study imaging of brain metabolism. Metabolism features include the amount of dopamine, gamma-aminobutyric acid, glutamate. Patients will be retested for PET after 6 months of implant.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, Study Chair — Shanghai Mental Health Center
Locations (2):
- China (2):
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No